CLINICAL TRIAL: NCT04935307
Title: Central Processing of Odour Stimuli in Patients With Multi-systemic Functional Somatic Disorder, Multiple Chemical Sensitivityor Post Covid Compared to Healthy Controls - the Pilot Study
Brief Title: Central Processing of Odour Stimuli in Patients With Functional Somatic Disorder, MCS or Post Covid Compared to Healthy Controls
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-273-20 MR pilot
Record Dates: First submitted 2021-06-09; First posted 2021-06-23 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Functional Disorder; Bodily Distress Syndrome; Multiple Chemical Sensitivity; Post COVID-19
MeSH Terms: conditions — Multiple Chemical Sensitivity | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: The aim of this study is to identify specific MRI and paraclinical measures for multiple chemical sensitivity (MCS), multi-organ bodily distress syndrome (multi-organ BDS) and post covid compared to Healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients with multiple chemical sensitivity (MCS) (Experimental): MCS is characterized by odour intolerance and various somatic symptoms attributed to the influence of toxic environmental chemicals in low usually harmless doses.
  Interventions: Diagnostic Test: MRI and paraclinical tests
- Patients with multi-systemic functional somatic disorders (FSD) (Experimental): Based on empirical research, a phenotype of multi-systemic FSD or multi-organ bodily distress syndrome (multi-organ BDS) has been identified in the most severely affected patients who have symptoms from multiple organ systems, thus fulfilling the criteria for multiple FSS. Multi-organ BDS is a research diagnosis, and the terms FSD and BDS are used as synonyms. This diagnosis is defined by an identifiable physical symptom pattern with symptoms from four groups (a cardiopulmonary, a gastrointestinal, a musculoskeletal, and a general symptom group).
  Interventions: Diagnostic Test: MRI and paraclinical tests
- Healthy controls (Experimental): Healthy participants
  Interventions: Diagnostic Test: MRI and paraclinical tests
- Patients with post-covid (Experimental): Post covid is according to WHO characterized by continuation og development of new symptom 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation. Symptoms include fatigue, shortness of breath and cognitive dysfunction over 200 different symptoms have been reported that can have an impact on everyday functioning.
  Interventions: Diagnostic Test: MRI and paraclinical tests

INTERVENTIONS:
Diagnostic Test: MRI and paraclinical tests — The patients and controls will be evaluated using MRI and furthermore a large test battery of questionnaires and paraclinical tests. Including the following test: MCS checklist, BDS-Checklist, Symptom Checklist-92 (SCL-92), Whiteley-8, SF-36, Major Depression Inventory (MDI), GAD-10 anxiety scale, and related questionnaire, behavioral olfactory test (TDI), habituation test, pain measurement thresholds tests, Heart Rate Variability and cognitive testing.

SUMMARY:
Background:

Functional somatic disorders (FSD) are frequent in all medical settings and characterized by persistent physical symptoms that cannot be explained by other somatic or psychiatric conditions. In recent decades, a number of different types of functional somatic disorders have been defined, but so far there is no clear explanation for the pathophysiology.

The high prevalence of olfactory problems in some patients with FSD suggests that olfactory symptoms are a potential diagnostic biomarker, especially in patients with multiple chemical sensitivity (MCS) and/ or post-covid.

The olfactory system is a unique sense with direct pathways to the limbic system, which is associated with emotion and mood. The focus on the olfactory system has revealed a significant association of this sense with numerous diseases.

Hypotheses:

* Patients with MCS and FSD have normal olfactory tests (normosmic subjects according to TDI score using "sniffing test") but differ in habituation test compared to healthy controls.
* MCS, post-covid and FSD patients have different odour perception processing in the brain as a "fingerprint" of functional somatic disorder compared to healthy controls.

Research plan:

The aim of this parts of the study is to identify specific MRI and paraclinical measures for MCS, post covid and BDS. In the first phase, 5 patients with MCS and 5 healthy controls will have a full clinical test of the olfactory system at the Flavour Institute, AU. In addition, they will be scanned (for "fingerprinting") where the investigators expect to find changes in olfactory connectivity similar to those seen in depression. This phase of the study will lead to a conclusion on the exact MR parameters to be used in the main study. In the second phase of the study, 10 patients with MCS, 10 with post-covid, 10 with FSD, and 10 healthy controls will be evaluated using a test battery of questionnaires and paraclinical tests.

Perspectives:

Previous imaging studies have focused on pain stimulation paradigms, rest-state fMRI, and DTI, but the olfactory system may be the "missing link" in identifiying a quantitative candidate in terms of whole-brain computational modeling and could potentially be used as a "fingerprint" in diagnosis and treatment monitoring.

DETAILED DESCRIPTION:
Background:

Functional somatic disorders (FSDs) are frequent in all medical settings and characterized by persistent physical symptoms that cannot be explained by other somatic or psychiatric conditions. Numerous terms have been used for the phenomenon, such as medically unexplained symptoms, somatoform disorders, and functional somatic syndromes (FSS). Various types of FSS exist, including chronic fatigue syndrome, myalgic encephalopathy, fibromyalgia, irritable bowel syndrome, and multiple chemical sensitivity (MCS), however previous studies suggest significant overlaps among most of them.

Based on empirical research, a phenotype of multi-systemic FSD or multi-organ bodily distress syndrome (multi-organ BDS) has been identified in the most severely affected patients who have symptoms from multiple organ systems, thus fulfilling the criteria for multiple FSS. Multi-organ BDS is a research diagnosis, and the terms FSD and BDS are used as synonyms. This diagnosis is defined by an identifiable physical symptom pattern with symptoms from four groups (a cardiopulmonary, a gastrointestinal, a musculoskeletal, and a general symptom group). The diagnosis has been included in the draft of WHO's ICD-11 for Primary Health Care under the name Bodily Stress Disorder. Multiple chemical sensitivity (MCS) is non-allergic and falls within the following two diagnostic categories: FSS and single-organ BDS. MCS is characterized by odour intolerance and various somatic symptoms attributed to the influence of toxic environmental chemicals in low usually harmless doses. Post-covid is charcterised by WHO by as continuation or development of new symptoms 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation. the symptoms includefatigue, shortness of breath and cognitive dysfunction over 200 different symptoms have been reported that can have an impact on everyday functioning.The studies conducted by Per Fink and colleagues in recent years imply a high prevalence of FSD (about 10%) in the Danish population, and that FSD is associated with severe individual and social consequences.

There is no clear explanation for the pathophysiology of FSD. Numerous hypotheses for the aetiology of FSD and MCS exist, including inflammation, immune system involvement, central sensitization, mental or physical lifelong stress, and hyperactivity of the autonomic nervous system, but recent studies raise a neurobiological basis in this issue. However, most neuroscientific studies lack generalizability due to a gap in the delimitation of FSD, which makes it difficult to treat FSDs adequately.

Hypotheses concerning odour intolerance include stressors of the olfactory system and immunological sensitization. Clinical observations indicate that hypersensitivity to olfactory stimuli is also at play in patients with BDS, and a study indicates that this also applies to patients with functional motor disorders.

The olfactory system is a unique sense with direct pathways to the limbic system that is associated with emotion and mood. Focus on the olfactory system has revealed significant associations between smell and neurodegenerative disorders, depression, schizophrenia, autism, ADHD, anorexia, addiction, trauma, and infections such as covid-19. At the moment, these associations can be used as a supportive diagnostic tool in Alzheimer's and Parkinson's disease as olfactory deficit signs are seen a few years before the onset of classic movement and cognition symptoms of these diseases.

The recent decade has seen the advent of the connectomics approach ("fingerprint"), a whole-brain analysis in neuroimaging, with considerable progress in mental illness. Currently, there are no method available to measure a potential central response to bodily sensations in patients with FSDs or to measure potential pathological processing of bodily stimuli in the brain. Until now, the focus has been on the pain or face stimulation paradigm.

The olfactory system may be the "missing link" for a quantitative candidate to differentiate patient groups on a whole-brain level and could potentially be used in the diagnosis of functional somatic disorders. On this background, the investigators carry out a study in MCS patients with specific symptoms from the olfactory system, and multi-organ BDS patients who have a variety of symptoms in general. To simplify the terms the investigators will divide the mentioned patient groups into MCS, BDS and compare these groups to Healthy controls (HC).

Hypotheses:

* Patients with MCS and BDS have normal olfactory tests (normosmic subjects according to TDI score using "sniffing test") but differ in habituation test compared to HC.
* MCS, post-covid and BDS patients have different odour perception processing in the brain as a "fingerprint" of functional somatic disorder compared to healthy controls.

Materials and methods:

For the purpose of finding as specific measures as possible for MCS and BDS, the study will be initiated by a pilot face both on MRI and paraclinincal parameter. First, Five MCS and five HC will have a full clinical test of the olfactory system at the Flavor Institute, AU. Furthermore, they will be MR scanned (for "fingerprinting") where the investigators expect to find changes in olfactory connectivity as investigators have seen in depression by Gleesborg et al in an ongoing study. This part of the study will lead to a conclusion on the exact MR parameters that will be used in the main study. Secondly, ten MCS, ten post-cpvid, ten BDS, and ten HC will be evaluated using a large test battery of questionnaires and paraclinical tests. Including the following test: MCS checklist, BDS-Checklist, Symptom Checklist-92 (SCL-92), Whiteley-8, SF-36, Major Depression Inventory (MDI), GAD-10 anxiety scale, and related questionnaire, behavioral olfactory test (TDI), habituation test, pain measurement thresholds tests, Heart Rate Variability and cognitive testing. Again for the purpose of finding a solid test battery for the main study.

Recruitment:

Patients with MCS will be recruited in the general population through advertisements e.g. on the MCS website. The diagnostic criteria for MCS are: a) at least two types of trigger exposure (e.g. perfume, tar), B) at least one symptom from the CNS (e.g. headache, dizziness), C) at least one symptom from either respiratory system (e.g. nose, mouth, and eyes are included) or skin, heart/chest, muscles/joints, bladder, stomach. Furthermore, their condition must have resulted in impairment of daily life (e.g. change of cleaning routine, choice of shops for shopping) and in either their social life (e.g. use of public transport, attendance at meetings and social events) or work life (e.g. sick leave from work, interrupted education). Duration of MCS diagnosis should be at least 6 months and fulfil the general inclusion criteria in the study and not fulfilling the criteria of multi-organ BDS.

Female BDS patients from the Research Clinic of Functional Disorders or the Pain Clinic, Aarhus University Hospital, Denmark who have suffered from multi-organ BDS for at least 6 months and fulfil the inclusion criteria and do not have any exclusion criteria will be invited to participate in the study.

Post-covid patient will be include from the post-covis clinic at Aarhus University Hospital, Aarhus, Denmark.

Healthy volunteers will be recruited though advertisements e.g. Aarhus university hospital.

Inclusion criteria (MCS, post-covid or BDS): 1) Female patients 18-70 years old. 2) Patients with moderate or severe MCS or post-covid and not multi-organ BDS 3) Patients with moderate or severe multi-organ BDS and not MCS or post-covid. 4) Symptoms present >6 months. 5) Written and verbal informed consent and letter of authority.

Exclusion criteria (MCS or BDS) before the beginning of the study; 1) Current sinonasal illness or upper respiratory tract allergy, 2) Serious or unstable medical illness (e.g. Apoplexy, Parkinson's, Alzheimer's disease, ischemic extremity pain, renal failure, liver failure, epilepsy, Raynaud´s phenomenon that is confirmed by medical history and, if possible, compared to medical records.3) Current and previous diagnosis of mania, bipolar disorder, psychosis, severe agitation, imminent deliria, current suicide risk, alcohol or drug dependence (ICD-10). Confirmed by psychiatric history and, if possible, compared to psychiatric or medical records. 4) Pregnancy and lactation.5) MR & MEG scanner incompatibility, assessed by an MR/MEG control questionnaire. After the beginning of the study; 1) MRI diagnosis of incidental pathologic findings; lesions, hemorrhage, etc.2) The onset of acute depression or serve anxiety. Relevant transference to treatment option should be initiated immediately. 3) Suicide risk (treatment will be initiated immediately).4) Pregnancy and lactation.5) The patient wishes to leave the study.5) The patient cannot co-operate during the examination.

The primary screening of all patients (MCS, post-covid or BDS) will be done through the telephone. At the first visit, all patients will have a medical and psychiatric anamnesis by diagnostic interviews using Schedules for Clinical Assessment in Neuropsychiatry (SCAN) interview, and a clinical examination (medical and neurological), which will be carried out by experienced physicians who have also been trained in the interview technique. Furthermore, patients will have verbal and written information about the study. Patients who give written and verbal informed consent and will be enrolled in the study. The healthy controls will go through the same procedures.

Measurements:

Functional symptoms and disabilities:

Selection of the MCS and multi-organ BDS patients by clinical and scan assessment, interview and medical examination. Furthermore, questionaries' found in the pilot study e.g. MCS checklist, BDS checklist etc.

Paraclinical tests:

Tests identified in the pilot study e.g. Cognitive testing, pain thresholds and HRV.

Olfactory tests:

The standardized psychophysical olfactory test, the "Sniffing Stick" test; will be performed on all three groups of participants before the scanning session. This battery of tests consists of odor threshold (T), discrimination (D), and identification (I) parts. The total score (TDI) was determined by the sum of the three scores (T+D+I).

Habituation test; In order to test the flexible hedonic evaluation of odors in MCS and BDS compare to healthy controls the investigators will carry out habituation tests. The evaluation task asks the participant to rate the odors pleasantness, all individuals responses will be arranged by Likert scale 1-5.

MRI scanning:

The investigators seek to employ whole-brain computational modeling based on MRI-derived functional and structural connectomes. The investigators will use the 3T MR Siemens® scanner that is situated at Aarhus University Hospital. A T1 structural image sequence will be run to obtain an image for later co-registration. After scanning data analyses including pre-processing, first-level analyses, and higher-level analyses will carry out.

Perspectives:

The methods of this study, integrative assessment, a statistical correlation between clinical diagnoses, behavioural tests, and neuroimaging 'fingerprints" could lead to the novel discovery of biomarkers for FSDs. Parallel to deepening our knowledge about the olfactory system, the investigators hope this study will open new horizons in extending the validity of new "fingerprints" in other FSDs. Further assessment of the correlation between neuroimaging findings and other analyses like genotyping, plasma factors measurement, will be explored in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Female patients and healthy controls 18-70 years old.
* Patients with moderate or severe MCS or multi-organ BDS or post-covid.
* Symptoms present >6 months.
* Written and verbal informed consent and letter of authority.

Exclusion Criteria:

1. Before the beginning of the study; Current sinonasal illness or upper respiratory tract allergy.

   Serious or unstable medical illness (e.g. Apoplexy, Parkinson's, Alzheimer's disease, ischemic extremity pain, renal failure, liver failure, epilepsy, and Raynaud's phenomenon) that is confirmed by medical history and, if possible, compared to medical records.

   Current and previous diagnosis of mania, bipolar disorder, psychosis, severe agitation, imminent deliria, current suicide risk, alcohol or drug dependence (ICD-10). Confirmed by psychiatric history and, if possible, compared to psychiatric or medical records.

   Pregnancy and lactation.

   MR & MEG scanner incompatibility, assessed by an MR/MEG control questionnaire.
2. After the beginning of the study;

MRI diagnosis of incidental pathologic findings; Lesions, Hemorrhage, etc.

The onset of acute depression or serve anxiety. Relevant transference to treatment option should be initiated immediately.

Suicide risk (treatment will be initiated immediately).

Pregnancy and lactation.

The patient wishes to leave the study.

The patient cannot co-operate during the examination.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
"Fingerprinting" | Through study completion, an average of 6 months
  The investigators seek to employ whole-brain computational modeling based on MRI-derived functional and structural connectomes. The investigators will use the 3T MR Siemens® scanner that is situated at Aarhus University Hospital. A T1 structural image sequence will be run to obtain an image for later co-registration. After scanning data analyses including pre-processing, first-level analyses, and higher-level analyses will carry out.
"Sniffing Stick test" | Through study completion, an average of 6 months.
  The standardized psychophysical olfactory test, the "Sniffing Stick" test; will be performed on all three groups of participants before the scanning session. This battery of tests consists of odor threshold (T), discrimination (D), and identification (I) parts. The total score (TDI) was determined by the sum of the three scores (T+D+I).
  Habituation test; In order to test the flexible hedonic evaluation of odors in MCS and BDS compare to healthy controls the investigators will carry out habituation tests. The evaluation task asks the participant to rate the odors pleasantness, all individuals responses will be arranged by Likert scale 1-5.

SECONDARY OUTCOMES:
Pain thresholds | Through study completion, an average of 3 months.
  Pressure pain thresholds by the pressure algometer and cold pressure test with ice water
Heart Rate Variability | Through study completion, an average of 6 months.
  Heart Rate Variability during rest and deep breathing
Cognitive testing | Through study completion, an average of 6 months.
  Participants' cognitive function will also be examined by a series of mental tests. For example, the participant is asked to connect 25 dots on a piece of paper as quickly as possible and in the correct order. Another example is that participants have to repeat a series of numbers from front to back.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Gormsen, PhD, Principal Investigator — Functional Disorders
Locations (1):
- The Research Clinic for Functional Disorders, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No